CLINICAL TRIAL: NCT02525081
Title: Effect of ACE-Inhibition on Microvascular Function in Women With Assessed Microvascular Dysfunction and No Obstructive Coronary Artery Disease
Brief Title: Effect of ACE-Inhibition on Microvascular Function in Women With Assessed Microvascular Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Marie Mide Michelsen, Medical Doctor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACIM
Record Dates: First submitted 2015-08-03; First posted 2015-08-17 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Microvascular Angina
Keywords: Microvascular Angina; therapy
MeSH Terms: conditions — Microvascular Angina | interventions — Ramipril; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACE-inhibitor (Experimental): In both the placebo and Ramipril group medication will start with either 2,5 mg (Blood Pressure<130) or 5 mg (Blood Pressure>130) daily. After 2-3 weeks the dose is doubled to 5 mg or 10 mg unless blood pressure is below 115 mmHg. If blood pressure continues to be higher than 115 mmHg for patients up titrated to 5 mg treatment dose will be doubled to 10 mg at the third visit.
  Patients taking a dose of
  * 2,5 mg will take a half tablet a day
  * 5 mg will take one whole tablet a day
  * 10 mg will take two tablets a day
  Interventions: Drug: Ramipril (ACE-inhibitor)
- Placebo (Placebo Comparator): In both the placebo and Ramipril group medication will start with either 2,5 mg (Blood Pressure<130) or 5 mg (Blood Pressure>130) daily. After 2-3 weeks the dose is doubled to 5 mg or 10 mg unless blood pressure is below 115 mmHg. If blood pressure continues to be higher than 115 mmHg for patients up titrated to 5 mg treatment dose will be doubled to 10 mg at the third visit.
  Patients taking a dose of
  * 2,5 mg will take a half tablet a day
  * 5 mg will take one whole tablet a day
  * 10 mg will take two tablets a day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ramipril (ACE-inhibitor) — up to 10 mg
  Other Names: Ramipril
  Arms: ACE-inhibitor
Drug: placebo — up to 10 mg
  Arms: Placebo

SUMMARY:
The aim of this study is to explore effects of long term treatment with ACE-inhibitor on the small vessel function assessed by coronary flow reserve (CFR) by transthoracic echocardiography and flow mediated dilation in normotensive patients with small vessel disease (CFR<2.2) and Angina Pectoris but no obstructive coronary artery disease.

DETAILED DESCRIPTION:
BACKGROUND Microvascular angina is proposed to be myocardial ischemia caused by microvascular dysfunction. When the microvasculature is dysfunctioning, blood flow in the coronary vessels does not increase sufficiently to meet oxygen demand leading to ischemia and pain. In the absence of stenosis of major coronary arteries, coronary flow reserve (CFR) reflects coronary microcirculation. Up to 50% of patients with angina and no obstructive coronary artery disease (CAD) have impaired CFR, which is a strong predictor of poor cardiovascular prognosis. Furthermore CFR has been shown to be associated with conventional risk factors; among these hypertension.

ACE-inhibitor treatment of patients with Angina Pectoris and/or essential hypertension and no stenosis on coronary angiogram improves CFR measured invasively by Doppler Guidewire or gas chromotography suggesting an effect of ACE inhibition on the microvasculature. Studies assessing the effect of ACE-inhibition in hypertensive and mild coronary artery disease patients with CFR assessed by positron emission tomography (PET) showed divergent results. One study showed an improvement on both resting and hyperaemic myocardial blood flow , another showed an increased myocardial perfusion reserve post treatment and a third failed to show any significant effect. If the effect seen on CFR is indirectly mediated via treatment of hypertension or if ACE-inhibition has a direct effect on the microvasculature continues to be uncertain in patients with microvascular angina. Some studies show an effect on CFR in both normotensive and hypertensive patients with microvascular angina whereas other studies only show an effect in hypertensive patients and not in normotensive. Treating patients with diabetes and a CFR>2.0 with ACE-inhibitor has also proven efficient in increasing CFR measured by transthoracic Doppler echocardiography (TTDE) supporting the theory that ACE-inhibition could have a direct effect on the microvasculature. In animal studies ACE-inhibition has shown capability of preventing adverse vascular remodelling dissociated to its blood pressure lowering effect. ACE inhibitor treatment is thought to be associated with vascular changes in CAD patients. However Clinical trials have shown discrepant results regarding reduction of hard endpoints with ACE inhibition in high-risk CAD patients. It remains unclear if ACE-inhibition has a direct effect on the microvasculature in normotensive patients with microvascular angina.

Endothelial dysfunction assessed by Flow-dependent endothelium-mediated dilation (FMD) is associated with cardiovascular risk factors and more prominent in women. FMD predicts long term cardiovascular events in healthy subjects. Treatment with most types of ACE-inhibitors improves FMD shown in studies with patients with syndrome X, coronary artery disease, and hypertension and in healthy elderly. However Enalapril treatment did not show an affect on FMD.

AIM The aim of this study is to explore effects of long term treatment with ACE-inhibitor on the microvasculature and endothelial function assessed by coronary flow reserve (CFR) by transthoracic echocardiography and flow mediated dilation (FMD) in normotensive patients with microvascular dysfunction (CFR<2.2) and Angina Pectoris but NO-CAD.

HYPOTHESIS ACE inhibitor treatment reverts microvascular remodelling and endothelial dysfunction in patients with microvascular dysfunction and Angina Pectoris but NO-CAD thereby improving microvascular function and reducing symptoms.

RESEARCH DESIGN The study is a randomised double-blinded interventional study. 72 patients with microvascular dysfunction assessed by TTDE as a CFR<2.2 are recruited from the iPower (ImProve diagnOsis and treatment of Women with angina pEctoris and micRovessel disease) cohort (women with angina but no obstructive CAD examined with TTDE CFR), Region Zealand. Patients with hypertension will be excluded from the study.

The patients will be randomised to group 1 or 2:

1. Group 1: Oral ACE-inhibitor for 6±1,5 months
2. Group 2: Oral matching placebo for 6±1,5 months Examinations and measurements will be performed at baseline and after 6±1,5 months. There are furthermore 2 possible blood pressure (BP)/kidney function control visits depending on how many up titrations of treatment medicine are necessary for the individual patient. Compliance calls and control of adverse events will be made every month and the patient can also contact us with any concern.

Participation in the study is 6±1,5 months. 24 hours before final measurements Ramipril treatment will be discontinued. Ramipril treatment will be add-on to usual treatment.

RANDOMIZATION PROCEDURE Patients will be randomized into 2 equal groups receiving either Ramipril or placebo. Randomization is done by the pharmacy (Glostrup Apotek). ACIM (Effect of ACE-Inhibition on Microvascular Function in Women with Assessed Microvascular Dysfunction) Id-numbers (ACIM1-72) are allocated equally to either placebo or Ramipril treatment using simple randomization.

Randomization is concealed in a document sealed in an opaque envelope and can only be revealed at the end of the study. For individual patients in occurrence of a serious adverse event the sponsor or investigator will contact the pharmacy to reveal medication type. The sealed envelope will be locked in a cabinet at the office of the sponsor.

The sponsor, investigator, research assistant and patients will have no knowledge of which randomization group the patients belong to Id-numbers (ACIM1-72) will be allocated to patients in a consecutive order.

TRIAL MEDICINE AND BLINDING Study medication will be prepared by the pharmacy (Glostrup Apotek) in a double-blinded manner. Medication will be delivered in bottles containing 50/100 x 5 mg placebo tablets or 5 mg Ramipril (Ramipril®, Hexal) and both bottle containers and tablets are indistinguishable. Tablets are produced with a pressure sensitive score notch and can be divided into equal halves. Bottle containers will be labelled with a study id-number ACIM1-ACIM72 (identification number/treatment number), the batch and/or code number to identify the contents and packaging operation, the name of the investigator Marie Michelsen/research assistant and mobile number, pharmaceutical dosage form, route of administration, quantity of dosage units, indication of use: "clinical trial", the storage conditions, period of use (expiry date) and warning label: "keep out of reach of children". The directions for use will be made to a leaflet according to individual dosage because of different final dosage after up titrations.

In both the placebo and Ramipril group medication will start with either 2,5 mg (BP<130) or 5 mg (BP>130) daily. After 2-3 weeks the dose is doubled to 5 mg or 10 mg unless blood pressure is below 115 mmHg. If blood pressure continues to be higher than 115 mmHg for patients up titrated to 5 mg treatment dose will be doubled to 10 mg at the third visit. Blood pressure and kidney function will be controlled at each visit (see fig. 1). If patients have symptoms of hypotension (dizziness, syncope or high pulse) treatment dose will be reduced and/or other blood pressure lowering treatment discontinued or if necessary Ramipril treatment discontinued.

If oral ACE-inhibitors are not tolerated treatment will be discontinued. Regarding exclusion for treatment discontinuation please see "withdrawal criteria".

Patients taking a dose of

* 2,5 mg will take a half tablet a day
* 5 mg will take one whole tablet a day
* 10 mg will take two tablets a day Patients will be up titrated in same manner independent of which medication they are on. For each study id-number medication for up titration is available. Patients will receive the appropriate amount of bottles according to uptitrated dose level (annex 1).

Patients will be up titrated and monitored by a research assistant so the investigator making the primary endpoint measure is unaware of the final treatment dose. In case of any adverse events/reactions or serious events/reactions the research assistant will confer with the sponsor or a project physician if necessary and not the investigator to avoid awareness of medication type for person obtaining primary endpoint. Only in case of a suspected serious reaction medication type will be unblinded by the sponsor or investigator by calling the pharmacy, Døgnåbent Glostrup Apotek, with patients id/cpr-number. Regarding exclusion for unblinding please see "withdrawal criteria".

Analysis of echocardiographic measurements for primary and secondary measurements will be made minimum 1 month after baseline and final visit so the investigator is unaware of blood pressure measurements during examinations.

Control of compliance will be made at visits and hereafter every month by patient structured open questions interviews (visits and telephone) Furthermore patients will make a diary every day of pill intake and any symptoms (potential adverse effects).

At the end of the study the patient will return used pill containers with remaining tablets within. These will be counted again to ensure medication compliance and accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Patients from an established cohort of patients with non obstructive coronary artery disease
* Microvascular dysfunction defined as a transthoracic echocardiography measured coronary flow reserve (CFR) < 2.2
* A good quality (quality index > 3) examination
* A blood pressure ≤ 150 at last visit in iPower
* Patients who are not in treatment for documented hypertension

Exclusion Criteria:

* Current treatment with ACE-inhibitors or Angiotensin II-antagonists
* Atrial fibrillation
* Pace-maker
* Allergy towards Ace-inhibitor, Ramipril ® or tool-medicine: Dipyridamole/adenosine, Nitro-glycerine or rescue medicine: Theophylline
* Baseline CFR >2.5 when entering ACIM-study.
* No episodes of chest pain within 6 months before inclusion
* Coronary angiography with significant stenotic lesions (>/=50%)
* Other cause of chest discomfort deemed highly likely
* Left ventricular ejection fraction below 45% assessed by echocardiography at baseline measurement
* Significant valvular heart disease (Definition: Verified in medical records after echocardiography. If the echocardiographer in this study suspects valvular heart disease, the patient is referred for expert evaluation and excluded from the study until valvular disease has been excluded. All definitions are taken from the guidelines of the Danish Society of Cardiology (DCS).

  * Haemodynamic significant Aortic Stenosis: Valve area < 1 cm2 or <0.6 cm2/m2 body surface area.
  * Severe aorta Regurgitation (AR): Vena contracta > 6 mm, Moderate/severe left ventricle (LV) volume load, ERO > 0.3 cm².
  * Mitral Stenosis (MS): Valve area < 2.5 cm2.
  * Severe Mitral Regurgitation (MR): effective regurgitant orifice > 0.4 cm², Moderate/severe LV-load, Vena contracta > 6 mm.
* Congenital heart disease or cardiomyopathy verified in medical records
* Significant co-morbidity with < 1 year expected survival: decision made by the person responsible for inclusion based on the patient interview and/or medical records.
* Severe chronic obstructive pulmonary disease with forced expiratory volume in 1 second (FEV1)<50% of predicted
* Severe asthma defined as asthma which requires treatment with high dose inhaled corticosteroids (ICS) plus a second controller (long acting β2 agonist (LABA), leukotriene modifier, theophylline or systemic corticosteroids) to prevent it from becoming uncontrolled or which remains uncontrolled despite this therapy."
* Previous verified myocardial infarction (Definition: verified in medical records, ST segment elevation myocardial infarction (STEMI) (ST segment elevation, elevated enzymes) or non-ST-segment elevation myocardial infarction (NSTEMI) (elevated enzymes, ECG changes/no ECG changes).
* Previous revascularization (Percutaneous Coronary Intervention or coronary artery bypass grafting)
* Elevated cardiac biomarkers: Troponin > 50 ng/l (high sensitive) or > 0.03 μg/l (4. generation), creatinin kinase myoglobin (CKMB) > 4.0 μg/l (women).
* ECG with verified ST-segment elevation
* Language- or other barrier to giving informed consent (for example mental ability to understand project)
* Travel distance: a distance to research hospital requiring more than 3 hours of travel
* Patient unwilling to participate (Low burden of symptoms, other illnesses, "Lack of energy", transport problems, anxiety because of the examination, other).
* No signed informed consent.
* Other (Pregnancy, significant psychiatric disorder)
* glomerular filtration rate < 50 mL/min/1,73 m2

Ages: 18 Years to 86 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in coronary flow reserve to after intervention | Patients are followed on average 6 months
  Coronary flow reserve is assessed by non-invasive Trans-Thoracic Doppler Echocardiography (TTDE)

SECONDARY OUTCOMES:
Change from baseline in Seattle Angina Questionnaire to after intervention | Patients are followed on average 6 months
  Evaluated by validated questionnaires: Seattle Angina Questionnaire
Change from baseline in Endothelial function to after intervention | Patients are followed on average 6 months
  Endothelial function is assessed by flow mediated dilation of the brachial artery by ultrasound
Change from baseline in Systolic function by speckle tracking strain to after intervention | Patients are followed on average 6 months
  strain assessed by speckle tracking echocardiography
Change from baseline in Roses questionnaire to after intervention | Patients are followed on average 6 months
  Evaluated by validated questionnaires: Roses Questionnaire
Change from baseline in Vital exhaustion questionnaire to after intervention | Patients are followed on average 6 months
  Evaluated by validated questionnaires: Vital exhaustion questionnaire
Change from baseline in International physical activity questionnaire (IPAQ) questionnaire to after intervention | Patients are followed on average 6 months
  Evaluated by validated questionnaires: IPAQ questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eva Prescott, professor, Study Director — Sponsor GmbH; Marie Michelsen, MD, Principal Investigator — Principal Investigator
Locations (1):
- Bispebjerg Hospital, Copenhagen NV, Denmark

REFERENCES:
- [Derived] Michelsen MM, Rask AB, Suhrs E, Raft KF, Host N, Prescott E. Effect of ACE-inhibition on coronary microvascular function and symptoms in normotensive women with microvascular angina: A randomized placebo-controlled trial. PLoS One. 2018 Jun 8;13(6):e0196962. doi: 10.1371/journal.pone.0196962. eCollection 2018. PMID 29883497